CLINICAL TRIAL: NCT06137651
Title: A Phase I/Ib Trial of Trotabresib (BMS-986378), an Oral BET Inhibitor) in Combination With Vinorelbine and Radiation Therapy in HER2+ Breast Cancer Patients With Central Nervous System Metastasis and Leptomeningeal Disease (CA076-1008)
Brief Title: Trotabresib in Combination With Vinorelbine and Radiation Therapy for the Treatment of HER2+ Breast Cancer With Central Nervous System or Leptomeningeal Metastasis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated by the sponsor
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 22C02; NCI-2023-08757 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00220214; NU 22C02 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Breast Carcinoma; Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Neoplasm in the Leptomeninges
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms; Meningeal Carcinomatosis | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (radiation therapy, trotabresib, vinorelbine) (Experimental): Patients CNS metastases or LMD undergo radiation therapy over 7 days in the absence of disease progression or unacceptable toxicity. Patients then receive trotabresib PO QD on days 1-4 and vinorelbine IV over 6-10 minutes on days 4, 11, and 18 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo MRI, CT, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Drug: Trotabresib; Drug: Vinorelbine
- Cohort S (surgery, trotabresib, vinorelbine) (Experimental): Patients who undergo tumor resection receive trotabresib PO QD on days 1-4 and vinorelbine IV on day 4. Patients then undergo standard of care surgery. Patients may undergo radiation therapy after surgery per standard of care. Patients may then receive trotabresib PO QD on days 1-4 and vinorelbine IV over 6-10 minutes on days 4, 11, and 18 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo MRI, CT, and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Procedure: Resection; Drug: Trotabresib; Drug: Vinorelbine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Resection — Undergo surgery
  Other Names: Surgical Resection
  Arms: Cohort S (surgery, trotabresib, vinorelbine)
Drug: Trotabresib — Given PO
  Other Names: 4-(2-(Cyclopropylmethoxy)-5-methylsulfonylphenyl)-2-methylisoquinolin-1-one; BET Inhibitor CC-90010; CC 90010; CC-90010; CC90010
Drug: Vinorelbine — Given IV
  Other Names: Dihydroxydeoxynorvinkaleukoblastine

SUMMARY:
This phase I/Ib trial tests the safety, side effects, and best dose of vinorelbine when given in combination with trotabresib in treating patients with HER2 positive breast cancer that has spread to the central nervous system or leptomeninges (metastasis). Cancer cells that make too much HER2 may grow more quickly and are more likely to spread to other parts of the body as metastases, including the central nervous system. Trotabresib is part of a family of drugs called BET inhibitors. Trotabresib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Vinorelbine is in a class of medications called vinca alkaloids. It works by slowing or stopping the growth of cancer cells in your body. Giving trotabresib and vinorelbine may increase in the anti-cancer activity of vinorelbine when used in combination with radiation (radiotherapy).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD) and recommended Phase II dose of trotabresib in combination with vinorelbine (VNR). (Phase I) II. To measure the progression free survival (PFS) from the date of first treatment of trotabresib to the date of first observation of progressive disease in both intracranial and extracranial sites in patients with brain metastases (BMs) and/or leptomeningeal disease (LMD). (Phase Ib [Expansion])

SECONDARY OBJECTIVES:

I. To establish the safety of trotabresib in combination with VNR, measured by the number of patients with adverse events. (Phase I) II. To assess the tolerance and toxicity profile of trotabresib in combination with VNR following RT in HER2+ breast cancer patients with central nervous system (CNS) metastasis. (Phase Ib [Expansion]) II. To measure the overall survival (OS) from the date of first treatment to the date of death from any cause. (Phase Ib [Expansion]) III. To evaluate the response rate (RECIST v. 1.1 and RANO-BM criteria) in patients with measurable disease. (Phase Ib [Expansion])

EXPLORATORY OBJECTIVES:

I. Disease monitoring using circulating tumor cells (CTCs) and circulating tumor DNA in peripheral blood and CSF. (Phase 1/1b) II. Expression of MZF1 and beta III tubulin in tumor tissue at baseline and during/after treatment when available. (Phase 1/1b) III. Evaluation of treatment response by metabolic positron emission tomography (PET) imaging using a novel 68Ga-HER2-nanobody (separate imaging protocol for select patients, pending future amendment to this trial for enrollment. (Phase 1/1b) IV. To estimate the concentrations of vinorelbine and trotabresib in central nervous system tissue (both in enhancing and non-enhancing parts). (Cohort S)

OUTLINE: This is a phase I dose-escalation study of vinorelbine followed by a phase Ib dose expansion study. Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients central nervous system (CNS) metastases or leptomeningeal disease (LMD) undergo radiation therapy over 7 days in the absence of disease progression or unacceptable toxicity. Patients then receive trotabresib orally (PO) once daily (QD) on days 1-4 and vinorelbine intravenously (IV) over 6-10 minutes on days 4, 11, and 18 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo magnetic resonance imaging (MRI), computed tomography (CT), and collection of blood samples throughout the trial.

COHORT S (PRE-SURGICAL COHORT): Patients who undergo tumor resection receive trotabresib PO QD on days 1-4 and vinorelbine IV on day 4. Patients then undergo standard of care surgery. Patients may undergo radiation therapy after surgery per standard of care. Patients may then receive trotabresib PO QD on days 1-4 and vinorelbine IV over 6-10 minutes on days 4, 11, and 18 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo MRI, CT, and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 6 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed diagnosis of HER2+ breast cancer. Patients may be immunohistochemistry (IHC) 3+ and/or fluorescence in situ hybridization (FISH) positive for HER2. IHC 2+ HER2 patients are eligible with reflex FISH-positive testing with the ratio ≥ 2.0. Alternatively, circulating tumor DNA testing positive for HER2 mutation is accepted for eligibility
* Patients must have newly diagnosed or progressive brain and/or leptomeningeal metastases, and a change in management and of treatment regimen is indicated. There is no limit on the number and types of prior systemic or intrathecal therapies
* Subjects must have an estimated life expectancy ≥ 3 months
* At registration, patients must have an interval of at least 2 weeks after the end of prior cytotoxic chemotherapy or immunotherapy or previous RT, one week from prior targeted small molecule drug treatment, interval of ≥ 4 weeks from prior bevacizumab or nitrosourea. At treatment start of trotabresib, there must be an interval of ≥ 4 weeks since last cytotoxic chemotherapy (6 weeks for prior nitrosourea) or immunotherapy

  * Note: Anti-HER2 directed treatment is allowed to continue, however, should be switched to trastuzumab before initiation of trotabresib. No washout period is required
* Patients must be age ≥ 18 years on the day of signing consent
* Patients must exhibit Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Leukocytes (WBC) ≥ 3,000/mcL or absolute neutrophil count (ANC) ≥ 1,500/mcL (within 14 days prior to registration)
* Hemoglobin (Hgb) ≥ 10 g/dL (within 14 days prior to registration)
* Platelets (PLT) ≥ 75,000/mcL (within 14 days prior to registration)
* Total bilirubin < 1.5 x upper limit of normal (ULN) (except patient with documented Gilbert's syndrome, ≤ 5 x ULN) (within 14 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 3 x institutional ULN (within 14 days prior to registration)
* Creatinine < 1.5x upper limit of normal (ULN) (within 14 days prior to registration)
* Patients must be able to swallow oral medication
* Patients must have recovered from the toxic effects of prior therapies (≤ Grade 1); however, persistent alopecia, or other toxicities not constituting a safety risk or being attributed to the tumor (e.g. neurological symptoms) based on investigator's judgement are not an exclusion criterion)
* Patients who are currently participating in or have participated in a study of an investigational agent or device must have discontinued the use of the investigational drug or device ≥ 4 weeks from registration on this study

  * Note: COVID-19 vaccination is allowed prior to and during study treatment
* Patients with a ventriculoperitoneal or ventriculoatrial shunt must have an on/off device in their shunt systems to be eligible for the study. Patients must be able to tolerate shunt closure for approximately 4 hours without development of clinical signs of increased intracranial pressure
* Patients must be able and willing to undergo research blood draws
* Patients must consent to retrieval of archival tissue or pretreatment tumor biopsy for research purposes if extra tissue is available
* The effects of trotabresib on the developing human fetus are unknown. Vinorelbineis known to be teratogenic causing birth defects and fetal loss in animals at concentrations which are below the human therapeutic dose range. For this reason, patients of child-bearing potential, patients with sperm-producing reproductive capacity and partners with child-bearing potential of patients with sperm-producing reproductive capacity much use contraception as specified below. Additionally, pregnant patients and patients that are nursing can not participate in this study because vinorelbine has the potential for teratogenic or abortifacient effects as described above. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vinorelbine, breastfeeding should be discontinued if the mother is treated with vinorelbine

  * A patient of childbearing potential (POCBP) is a person who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy or other medical condition does not rule out childbearing potential) for at least 12 consecutive months and verified by an FSH blood test at screening. FSH test should be >30 mIU/mL but FSH will be low if the subject is taking hormone replacement therapy or oral contraceptives. The requirement for FSH testing may be waived for subjects greater than 62 years of age
* Patients of childbearing potential (POCBP) must:

  * Either commit to true abstinence from heterosexual intercourse (which must be reviewed monthly and source documented) or to use one highly effective contraceptive method. True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception). Highly effective contraceptive methods are combined (containing estrogen and progestogen) or progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, intravaginal, patch, or implantable); bilateral tubal ligation; intra-uterine device; intrauterine hormone-releasing system; or vasectomized partner sterilization (note that vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the POCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success). These measures should be used from 28 days before the first dose of study medication, throughout the study, and for 7 months following the last dose of trotabresib and 6 months after the last dose of vinorelbine, whichever is longer
  * Oocyte donations and nursing are prohibited during the same time period when highly effective contraception is required. Should a patient of child bearing potential experience a change in contraception method or become pregnant or suspect they are pregnant during the time period when highly effective contraception is required, they should notify the investigator immediately
  * Patients of child-bearing potential must have two negative serum or urine pregnancy tests (beta-subunit of human chorionic gonadotropin or beta-human chorionic gonadotropin [hCG]) as verified by the investigator prior to starting the study drugs. The second test should be performed on Day -1 or Day 1 prior to dosing. The pregnancy test (serum or urine) should have a sensitivity of at least 25 mIU/ml. Patients of child-bearing potential must agree to ongoing pregnancy testing monthly during dosing and for the same time period when highly effective contraception is required
* Patients with sperm-producing capacity must agree to contraception use as indicated below:

  * Patient with sperm-producing capacity condom use
  * Patients with sperm-producing capacity must practice true abstinence (which must be reviewed on a monthly basis) or agree to use a condom (a latex or non-latex synthetic condom is required) during any sexual activity (eg, vaginal, anal, oral) with a pregnant or nursing person or a person of child-bearing potential and will avoid conceiving from signing the informed consent form, while participating in the study, during dose interruptions, and for at least 4 months after the last dose of trotabresib or 6 months after the last dose of VNB, whichever is longer, even if they have undergone a successful vasectomy. Patients with sperm-producing capacity should inform the investigator immediately if they believes that their partner has become pregnant
  * Patients with sperm-producing capacity should not donate sperm for the same period of time that is required for condom use. Partners who are of child-bearing potential must use one highly effective form of contraception during the same time period that the patients with sperm-producing capacity must use a condom
* Patients must have the ability to understand and the willingness to sign a written informed consent document. Consent must be signed prior to registration on this study
* Cohort S only: Patient must be a candidate for a planned surgical resection of at least one central nervous system (CNS) metastasis, with an indication for surgical resection (e.g. mass effect, therapeutic intent in oligometastatic disease, diagnostic confirmation/determination of histologic and/or molecular tumor characteristics)
* Phase I/Ib only: Patients must have evaluable metastatic disease in the CNS and/or evidence of leptomeningeal disease (LMD) (clinically, on imaging or detected by circulating tumor cells)
* Phase I/Ib only: Patients must have unequivocal evidence of new and/or progressive brain metastases, and at least one of the following scenarios:

  * Prior treatment with Stereotactic radiosurgery (SRS ) or surgery, and residual surgically or radiosurgically un-treated lesions remaining. Such participants are eligible for immediate enrollment on this study providing that at least one untreated lesion is evaluable or measurable
  * Patients who have not previously been treated with cranial irradiation are eligible to enter the study
  * Patients are eligible independent of presence or absence of progressive systemic disease
* Phase I/Ib only: Patients must have an indication for local CNS-directed therapy, e.g. new metastases amenanble for radiotherapy or SRS, reduction of mass effect and/or palliation of symptoms
* Phase I/Ib only: Patients planned radiotherapy needs to be prescribed in accordance to generally acceptable guidelines and practice, i.e.:

  * Patients who have received prior whole brain radiotherapy should only be treated with stereotactic radiosurgery (SRS)
  * A delay of ≥ 3 months should be observed between prior whole-brain radiotherapy (WBRT) and SRS
  * Repeat SRS to a lesion previously treated with SRS is not allowed
  * There is no limit to the number of lesions that have previously bee treated with SRS, and there is no limit to the number of lesions to be treated with SRS, if clinically indicated

Exclusion Criteria:

* Patients who are on escalating doses of corticosteroids

  * Note: Patients must be on a stable or decreasing dose of corticosteroids equivalent to dexamethasone ≤ 8mg averaged over the last 7 days to be eligible for the study
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to trotabresib and vinorelbine (VNR)
* Patients who have a known additional malignancy that is progressing or requires active treatment

  * Note: Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Patients who have impaired cardiac function or clinically significant cardiac diseases, including any of the following:

  * LVEF < 45% as determined from review of any standard of care echocardiograms (ECHOs) multigated acquisition scans/(MUGAs) completed in the past 2 years
  * Complete left bundle branch or bifascicular block (verified by review of medical records)
  * Congenital long QT syndrome (verified by review of medical records)
  * Persistent or clinically meaningful ventricular arrhythmias or atrial fibrillation (verified by review of medical records)
  * Fridericia's correction formula (QTcF) ≥ 480 msec on screening electrocardiogram (ECG)
  * Unstable angina pectoris or myocardial infarction ≤ 6 months prior to starting therapy (verified by review of medical records)
* Patients who require ongoing treatment with chronic, therapeutic dosing of anti-coagulants (ex. warfarin, low molecular weight heparin, Factor Xa inhibitors, thrombin antagonists)

  * Note: Low dose low molecular weight heparin for catheter maintenance and for prophylactic use are permitted if medically indicated
* Patients who have a history of bleeding diathesis
* Patients who have any hemorrhage/bleeding event > Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or hemoptysis > 1 tsp within 4 weeks prior to treatment initiation
* Patients who have known prior episodes of non-arteritic anterior ischemic optic neuropathy should be excluded from the study

  * Note: Trotabresib should be used with caution in patients with retinitis pigmentosa. The Principal Investigator may be consulted
* Patients who have poor bone marrow reserve as indicated by the following scenarios:

  * Have received extensive bone radiotherapy
  * Have experienced several episodes of bone marrow aplasia in previous treatments
  * Confirmed histological bone marrow cancer infiltration
  * Require regular hematopoietic support with blood transfusions, erythropoietin or growth factors
* Patients who have an active infection requiring systemic therapy
* Patients who have had a major surgical procedure or significant traumatic injury within 21 days prior to day 1 of treatment on study

  * Note: Ommaya/programmable shunt placement is allowed
* Patients who have current evidence of any condition, therapy or laboratory abnormality that might confound the results of the trial, interfere with their participation for the full duration of the trial or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Patients who have a psychiatric illness/social situations that would limit compliance with study requirements
* Female patients who are pregnant or nursing. Pregnant women are excluded from this study because vinorelbine has the potential for teratogenic or abortifacient effects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (Phase I) | Up to 28 days after treatment
Incidence of adverse events (Phase Ib) | Up to 30 days after last dose
  To assess the toxicity profile of vinorelbine and trotabresib this endpoint will collect and report the frequency of adverse events by type, severity (grade), timing, and attribution to vinorelbine and trotabresib, according the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Toxicities will be summarized by maximum grade and patients with and without leptomeningeal spread will be evaluated separately.

SECONDARY OUTCOMES:
Incidence of adverse events (Phase I) | Up to 30 days after last dose
  To assess the toxicity profile of VNR and trotabresib this endpoint will collect and report the frequency of adverse events by type, severity (grade), timing, and attribution to VNR and trotabresib, according the NCI-CTCAE version 5.0. Toxicities will be summarized by maximum grade.
Progression-free survival (PFS) (Phase Ib) | Time that elapses between the initiation of trial therapy (cycle 1 day 1 [C1D1]) and the day of first documented disease progression or death from any cause for all evaluable patients, assessed up to 1 year
  Median PFS will be calculated based on the Kaplan-Meier estimates of PFS. PFS data will be collected from the initiation of trial therapy (C1D1) until the patient experiences disease progression, initiates subsequent anti-cancer therapy, completes study participation, or experiences death from any cause (whichever is sooner). If disease progression or death from any cause is not observed prior to initiating subsequent anti-cancer therapy or completing study participation, the PFS will be censored as the last available disease assessment.
Overall survival (OS) (Phase Ib) | Time that elapses between the initiation of trial therapy (C1D1) and the date of death from any cause for all evaluable patients, assessed up to 1 year
  Medium OS (mOS) will be calculated based on the Kaplan-Meier estimates of OS. OS data will be collected from the initiation of trial therapy (C1D1) until the patient completes study follow up participation, experiences death from any cause or is documented as lost to follow up per institutional standard (whichever is sooner). If death from any cause is not observed prior to completing study participation, the OS will be censored as the time of the last available documentation of survival status. Last available documentation of survival status is defined as the date of death or the latest of the following times: treatment discontinuation date, last dosing administration date, last disease assessment date, or the last follow-up date when the patient was known to be alive.
Objective response rate (ORR) (Phase Ib) | Time that elapses between the initiation of trial therapy (C1D1) and the date of death from any cause for all evaluable patients, assessed up to 1 year
  will calculate the proportion of treated patients who experience an objective response [confirmed complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.11 and Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) criteria. Confirmation of response should be conducted via imaging ≥ 28 days after the response was first documented. The date of first response for either CR or PR will be used for the calculation of ORR. ORR data will be collected from the initiation of trial therapy (C1D1) until the response has been confirmed, the patient experiences disease progression, initiates subsequent anti-cancer therapy, or completes study participation (whichever occurs first). Will also determine the objective response rate specifically for intracranial/central nervous system (CNS) disease, disease sites with and without radiotherapy, and extracranial disease.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Stupp, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States